CLINICAL TRIAL: NCT06958718
Title: Efficacy of Ultrasound-guided Versus Surgical Erector Spinae Plane Block With a Mixture of Bupivacaine and Dexmedetomidine in Lumbar Spinal Fusion Surgery: A Prospective Randomized Double-Blinded Clinical Trial.
Brief Title: Ultrasound vs. Surgical ESP Block With Bupivacaine-Dexmedetomidine in Lumbar Fusion Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Associate Professor of Anesthesiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: M762
Record Dates: First submitted 2025-04-21; First posted 2025-05-06 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Post Operative Pain
Keywords: lumbar spinal surgery; Pain; ESPB; Ultrasound guided ESPB; Surgical ESPB; Dexmedetomidine
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Guided erector spinae plane block (UB) (Active Comparator): the block will be done using ultrasound device after wound closure
  Interventions: Procedure: Ultrasound Guided erector spinae plane block (UB); Drug: Dexmedetomidine; Drug: Bupivacaine Hcl 0.5% Inj
- Surgical erector spinae plane block (SB) (Active Comparator): the block will be done surgically before wound closure
  Interventions: Procedure: Surgical erector spinae plane block (SB); Drug: Dexmedetomidine; Drug: Bupivacaine Hcl 0.5% Inj

INTERVENTIONS:
Procedure: Ultrasound Guided erector spinae plane block (UB) — Ultrasound Guided erector spinae plane block (UB) with 40 ml Bupivacaine HCL mixed with 0.5 μg/kg dexmedetomidine .. After the surgical incision is closed and before extubation, while the patient remains in the prone position. A linear high-frequency transducer (L6-12 linear array transducer (6-12 MHz) on GE Healthcare logiq p7, made in Korea) will be positioned in a sagittal orientation, 4 cm lateral to the L3 transverse process. A 22 G × 88 mm block needle will be inserted in the craniocaudal direction, with the needle tip placed beneath the erector spinae muscle and above the hyperechoic transverse process. The needle tip position will be confirmed via saline injection. Once correct needle placement is verified, 40 mL of 0.25% bupivacaine, combined with 0.5 μg/kg dexmedetomidine 15 will be administered divided on both sides.
  Arms: Ultrasound Guided erector spinae plane block (UB)
Procedure: Surgical erector spinae plane block (SB) — Surgical erector spinae plane block (SB) with 40 ml Bupivacaine HCL mixed with 0.5 μg/kg dexmedetomidine ..This volume will be divided into 8 injections, four 5 ml injections on each side. The surgeons will perform the block just before starting the wound closure stage. The surgical ESP block technique consists of injections at four bilateral levels, starting from one level above the operated vertebra and covering all surgical segments using a 22G × 88 mm needle. The needle will be inserted to contact the transverse process, and the injectate will be delivered between the erector spinae muscle and the transverse process at each level.
  Arms: Surgical erector spinae plane block (SB)
Drug: Dexmedetomidine — 0.5 μg/kg dexmedetomidine added to block solution
  Other Names: precedex
Drug: Bupivacaine Hcl 0.5% Inj — 40 ml Bupivacaine HCL
  Other Names: Marcaine

SUMMARY:
Lumbar spine surgery causes intense post-op pain, peaking within 12 hours and improving by day three. Traditional spinal procedures involve extensive tissue dissection, leading to severe pain and potential complications like delayed mobilization, respiratory issues, and chronic pain. Effective pain management is crucial. Opioid-based relief is standard but comes with side effects (nausea, respiratory depression), increasing hospital stays and costs.

Dexmedetomidine (DEX) is an alpha-2 adrenergic receptor agonist that enhances nerve block duration when combined with local anesthetics (LAs). It works by inhibiting sodium and potassium channels, leading to prolonged hyperpolarization.

Regional nerve blocks, such as thoracic epidurals and fascial plane blocks, improve postoperative pain management and help reduce opioid use, minimizing complications. Various techniques, including ESP blocks, paravertebral Block (PVB), and Serratus anterior Block (SAB) have been explored for acute pain relief.

The Erector Spinae Plane Block (ESPB), initially used for thoracic neuropathic pain, has expanded to thoracic, breast, and abdominal surgeries.

The ESP block is done by injecting a local anesthetic between the transverse process and the erector spinae muscle. Ultrasound guidance helps visualize the spread of the anesthetic and the surrounding anatomy. Previous studies indicate that the ESP block can effectively relieve pain after lumbar spine surgery and may reduce postoperative opioid use when local anesthetics are applied to the wound and deep tissues. Based on this, performing the ESP block directly by the surgical team, using a local anesthetic between the erector spinae muscle and transverse process with direct view and free hand, may yield similar results to the ultrasound guided technique. The current study aims to evaluate the analgesic efficacy of Ultrasound-Guided Erector Spinae Plane Block in comparison with surgical Erector Spinae Plane Block using a mixture of bupivacaine and dexmedetomidine in lumbar Spinal fusion Surgeries.

DETAILED DESCRIPTION:
After approval of the local institutional ethics committee and local institutional review board. Patients scheduled for elective lumbar spinal Fusion surgeries and fulfilling the inclusion criteria in Fayoum University Hospital starting from February 2025 will be enrolled in this prospective randomized study until fulfilling the sample size. The eligible participants will sign a detailed informed consent before recruitment.

Randomization will be done using computer-generated random numbers placed in separate opaque envelopes and opened by the anesthesiologist just before induction of anesthesia, eligible patients will be randomized with 1:1 allocation ratio into two groups:

* The surgical ESPB group (SB)
* The Ultrasound guided ESPB group (UB) Both the anesthesiologist and the surgeons performing the US guided ESP block and surgical ESP block will not be further involved in the study. Another anesthesiologist will be responsible for further patient care and data collection. This anesthesiologist and the patient will be blinded from the group assignments.

General anesthesia:

Upon arrival at the operating theatre, all patients will be monitored using electrocardiography, pulse-oximetry, capnography, and Noninvasive blood pressure (NIBP). After routine history, examination, and review of laboratory results, General anesthesia will be induced with intravenous propofol (2 mg/kg), fentanyl (1 μg/kg), and atracurium (0.5mg/kg). After that, patients will be intubated and placed in a prone position. Anesthesia will be maintained using IV atracurium and inhalational anesthesia (isoflurane) in an oxygen and fresh air mixture. All patients will receive intravenous Ketorolac (30 mg), Nalbuphine (10 mg), and Ondansetron 8 mg approximately 30 min before the end of the surgery.

Block technique:

For patients in Group UB, an ultrasound-guided ESP block will be performed after the surgical incision is closed and before extubation, while the patient remains in the prone position. A linear high-frequency transducer (L6-12 linear array transducer (6-12 MHz) on GE Healthcare logiq p7, made in Korea) will be positioned in a sagittal orientation, 4 cm lateral to the L3 transverse process. A 22 G × 88 mm block needle will be inserted in the craniocaudal direction, with the needle tip placed beneath the erector spinae muscle and above the hyperechoic transverse process. The needle tip position will be confirmed via saline injection. Once correct needle placement is verified, 40 mL of 0.25% bupivacaine, combined with 0.5 μg/kg dexmedetomidine 15 will be administered divided on both sides. For patients in group SB, the injectate will be prepared with the help of the anesthetist by adding 0.5 μg/kg dexmedetomidine to 40 mL of 0.25% bupivacaine. This volume will be divided into 8 injections, four 5 ml injections on each side. The surgeons will perform the block just before starting the wound closure stage. The surgical ESP block technique consists of injections at four bilateral levels, starting from one level above the operated vertebra and covering all surgical segments using a 22G × 88 mm needle. The needle will be inserted to contact the transverse process, and the injectate will be delivered between the erector spinae muscle and the transverse process at each level.

Postoperative pain management:

After discharge to ward, all patients will receive paracetamol 1g / 8hrs, ketorolac 30 mg/ 12hrs and nalbuphine 5mg as a rescue analgesia. The patient's pain will be evaluated using a Visual Analog Scale (VAS) where 0 denotes no pain, and 10 represents the most intense pain ever experienced. Dynamic and static VAS scores will be recorded in the postoperative period at 1, 4, 8, 16, 24, 36 and 48 hours. Patients with VAS scores of 4 or higher will receive Nalbuphine (5 mg) for rescue analgesia.

sample size calculation and statistical analysis : Sample size was calculated using IBM SPSS 29 software for windows (IBM Co., Armonk, NY, USA). Calculation of the sample size was based on the ability to detect a difference of one point in the VAS score between the two groups based on the results of a study by Kaciroglu, A. et al. At least 23 patients are needed per group to detect this difference at α level of 0.05 and study power of 80%. We decided to recruit 26 patients per group to compensate for any possible withdrawals up to 10% and to increase the study power. The sample size calculation was based on the independent samples t test. Statistical analysis will be performed using SPSS for Windows, version 29 (IBM Corp., and Armonk, New York, USA). Descriptive statistics will be presented in the form of (mean ± SD), or (median with interquartile range) for numerical data, while numbers and percentages will be used for categorical data. Testing for normality of distribution will be done using the Shapiro-Wilk test. Categorical variables will be analyzed using Chi-square test or Fisher's exact test. Differences in parametric normally distributed numerical data will be compared using Student's t tests, While the non-parametric data will be compared using Mann Whitney U-test. Results will be considered statistically significant if the p value is less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

- American Society of Anesthesiologists (ASA) I-Ⅲ patients scheduled for elective two or three levels of lumbar spinal fusion surgeries by the same surgical team.

Exclusion Criteria:

* Patient refusal.
* Body mass index > 30 kg/m2
* Significant renal, hepatic, or cardiovascular diseases.
* History of allergy to one of the study drugs (local anesthetics, opioids, or dexmedetomidine).
* Any contraindications to regional anesthesia like local infection or abnormal coagulation function.
* Pregnant or breastfeeding women.
* Chronic opioid use, history of chronic pain, or cognitive disorders.
* Emergent surgeries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
QAQStatic VAS score one hour postoperatively. | one hour after surgery
  Visual Analog Scale (VAS) tool used to measure pain of patients after surgery, consist of 100mm length scale where 0 = "no pain" and 100 = "worst imaginable pain". static VAS score to be obtained one hour after surgery.

SECONDARY OUTCOMES:
Postoperative static VAS scores. | At 48 hours after the block
  Visual Analog Scale (VAS) tool used to measure pain of patients after surgery, consist of 100mm length scale where 0 = "no pain" and 100 = "worst imaginable pain". static VAS score to be obtained at 2, 4, 8, 16, 24, 36, and 48 hours after the block.
Postoperative dynamic VAS scores. | At 48 hours after the block
  Visual Analog Scale (VAS) tool used to measure pain of patients after surgery, consist of 100mm length scale where 0 = "no pain" and 100 = "worst imaginable pain". Dynamic VAS score to be obtained at 2, 4, 8, 16, 24, 36, and 48 hours after the block.
Time consumed in the block. | the time After starting blocking procedure till finishing procedure up to 1 hour
  Time of the block procedure
The time of the first postoperative analgesic request. | the time After blocking procedure till the first request of analgesia up to 48 hours
  The time consumed after block until first request of analgesia.
Total postoperative needs of nalbuphine. | At first 24 hours after ESP block.
  amount of nalbuphine used in milligrams.
Heart rate (HR) | Assessed up to 48 hours after block.
  at 0 (block time), 5min, 10 min, 15 min, 30 min, 1h, 2h, 4h, 8h, 16h, 24h, 36h, and 48h after ESP block.
Mean Arterial Pressure (MAP) | Assessed up to 48 hours after block.
  at 0 (block time), 5min, 10 min, 15 min, 30 min, 1h, 2h, 4h, 8h, 16h, 24h, 36h, and 48h after ESP block.
number of participants with nausea and vomiting. | Assessed up to 48 hours after block.
  Complications related to the block or study medications.
Incidence of respiratory depression | At first 24 hours after ESP block.
  Respiratory Rate < 8 bpm.
number of participants with pruritus | At first 24 hours after ESP block.
  Complications related to the block or study medications
number of participants with manifestations of systemic toxicity from local anesthetic drugs | At first 24 hours after ESP block.
  Assess for neurological or cardiovascular toxicity symptoms
Sedation level | Assessed up to 24 hours after block.
  Assess sedation level, using a four-point sedation scale (score 1 = spontaneous eye opening [awake and alert]; score 2 = drowsy, responsive to verbal stimuli.
  score 3 = drowsy, arousable to physical stimuli; score 4 = unresponsive) ِِAssessed at 1, 2, 4, 8, 16, 24 hours after the block
24h Quality of recovery questionnaire (QoR-15) | 24 hours after surgery.
  15 items questionnaire used to evaluate the quality of recovery 24h after surgery, an aggregate score from 0 (no recovery) to 150 (total recovery)
Length of hospital stay | The Time of stay (surgery day) until hospital discharge up to 7 days
  measured in days, from day 0, the day of surgery, until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Hamed, MD, Principal Investigator — Fayoum University Hospital; Mohamed A Elsaeed, MD, Study Director — Fayoum University Hospital
Locations (1):
- Fayoum University hospital, Al Fayyum, Fayoum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kleif J, Gogenur I. Severity classification of the quality of recovery-15 score-An observational study. J Surg Res. 2018 May;225:101-107. doi: 10.1016/j.jss.2017.12.040. Epub 2018 Feb 21. PMID 29605019
- [Background] Kraiwattanapong C, Arnuntasupakul V, Kantawan R, Woratanarat P, Keorochana G, Langsanam N. Effect of Multimodal Drugs Infiltration on Postoperative Pain in Split Laminectomy of Lumbar Spine: A Randomized Controlled Trial. Spine (Phila Pa 1976). 2020 Dec 15;45(24):1687-1695. doi: 10.1097/BRS.0000000000003679. PMID 32890299
- [Background] Singh S, Choudhary NK, Lalin D, Verma VK. Bilateral Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia in Lumbar Spine Surgery: A Randomized Control Trial. J Neurosurg Anesthesiol. 2020 Oct;32(4):330-334. doi: 10.1097/ANA.0000000000000603. PMID 31033625
- [Background] Devin CJ, McGirt MJ. Best evidence in multimodal pain management in spine surgery and means of assessing postoperative pain and functional outcomes. J Clin Neurosci. 2015 Jun;22(6):930-8. doi: 10.1016/j.jocn.2015.01.003. Epub 2015 Mar 9. PMID 25766366
- [Background] Qiu Y, Zhang TJ, Hua Z. Erector Spinae Plane Block for Lumbar Spinal Surgery: A Systematic Review. J Pain Res. 2020 Jul 1;13:1611-1619. doi: 10.2147/JPR.S256205. eCollection 2020. PMID 32669870
- [Background] Liang X, Zhou W, Fan Y. Erector spinae plane block for spinal surgery: a systematic review and meta-analysis. Korean J Pain. 2021 Oct 1;34(4):487-500. doi: 10.3344/kjp.2021.34.4.487. PMID 34593667
- [Background] Chitnis SS, Tang R, Mariano ER. The role of regional analgesia in personalized postoperative pain management. Korean J Anesthesiol. 2020 Oct;73(5):363-371. doi: 10.4097/kja.20323. Epub 2020 Aug 5. PMID 32752602
- [Background] Bajwa S, Kulshrestha A. Dexmedetomidine: an adjuvant making large inroads into clinical practice. Ann Med Health Sci Res. 2013 Oct;3(4):475-83. doi: 10.4103/2141-9248.122044. PMID 24379995
- [Background] Prabhakar NK, Chadwick AL, Nwaneshiudu C, Aggarwal A, Salmasi V, Lii TR, Hah JM. Management of Postoperative Pain in Patients Following Spine Surgery: A Narrative Review. Int J Gen Med. 2022 May 2;15:4535-4549. doi: 10.2147/IJGM.S292698. eCollection 2022. PMID 35528286
- [Background] Bianconi M, Ferraro L, Ricci R, Zanoli G, Antonelli T, Giulia B, Guberti A, Massari L. The pharmacokinetics and efficacy of ropivacaine continuous wound instillation after spine fusion surgery. Anesth Analg. 2004 Jan;98(1):166-172. doi: 10.1213/01.ANE.0000093310.47375.44. PMID 14693613